CLINICAL TRIAL: NCT01789086
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess Safety, Tolerability and Pharmacokinetics of Liraglutide in Obese Adolescent Subjects Aged 12 to 17 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-3967; 2012-000038-20 (EudraCT Number); U1111-1126-8119 (Other: WHO)
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Administered subcutaneously (s.c., under skin) for 5-6 weeks. Initial dose of 0.6 mg/day. The dose will be escalated by 0.6 mg/day in weekly steps to a maximum of 3.0 mg/day
  Arms: Liraglutide
Drug: placebo — Administered subcutaneously (s.c., under skin) for 5-6 weeks. Initial dose of 0.6 mg/day. The dose will be escalated by 0.6 mg/day in weekly steps to a maximum of 3.0 mg/day
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The purpose of the trial is to assess safety, tolerability and pharmacokinetics (the exposure of the trial drug in the body) of liraglutide in obese adolescent subjects aged 12 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Tanner stage 2-5 pubertal development at time of randomisation
* Body Mass Index (BMI) corresponding to 30 kg/m^2 or above for adults by international cut-off points and 45 kg/m^2 or below and equal to or above 95th percentile for age and gender
* Fasting plasma glucose below 7.0 mmol/L (126 mg/dL) (central laboratory analysis)

Exclusion Criteria:

* Subjects with clinically diagnosed secondary causes of childhood obesity such as chromosomal abnormalities (e.g. Turner syndrome), syndromic obesity (e.g. Prader Willi syndrome) or endocrinologic disorders (e.g. Cushing Syndrome)
* Subjects with confirmed diagnosis of bulimia
* Subjects with Tanner stage 1 development (prepubertal)
* Diagnosis of type 1 or type 2 diabetes mellitus as judged by the investigator
* Previous treatment with a GLP-1 (glucagon-like peptide 1) receptor agonists (e.g. exenatide or liraglutide or other), DPP-4 (dipeptidyl peptidase-4) inhibitors, orlistat or other weight lowering medication, any antipsychotic medication or systemic corticosteroids within the last 3 months
* Currently using or have used within 3 months before screening for this trial: any systemic treatment that in the opinion of the investigator interferes with PK (pharmacokinetic), PD (pharmacodynamic) and safety endpoints
* Surgical treatment for obesity
* Past or current chronic or idiopathic pancreatitis, or any of the following: -amylase or lipase above 2 times UNR (upper normal range), -triglycerides above 500 mg/dL, -calcium above UNR, -history of gallstones (not treated by cholecystectomy)
* Uncontrolled treated or untreated hypertension 99th percentile for age and gender in children
* History of major depressive disorder or history of other severe psychiatric disorders (e.g. schizophrenia or bipolar disorder) that could in the opinion of the investigator interfere with trial compliance or subject safety
* Subjects with a history of suicide attempts or history of any suicidal behaviour within the past month before entry into the trial

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From the time of first dosing (Day 0) and until completion of follow-up visit (up to 6 weeks' treatment and 5-14 days subsequent follow-up period)

SECONDARY OUTCOMES:
Incidence of liraglutide antibody | At follow-up (up to 6 weeks' treatment and 5-14 days subsequent follow-up period)
At steady state at each dose step: C-trough | After 7, 14, 21, 28 and 35 days of treatment
At steady-state: model-derived area under the liraglutide concentration curve over the dosing | Last dose day, after up to 6 weeks' treatment
At steady-state: model-derived t½ (terminal half-life) | Last dose day, after up to 6 weeks' treatment
At steady-state: model-derived CL/F (apparent clearance) | Last dose day, after up to 6 weeks' treatment
At steady-state: model-derived V/F (apparent volume of distribution) | Last dose day, after up to 6 weeks' treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hanover, Germany

REFERENCES:
- [Result] Danne T, Biester T, Kapitzke K, Jacobsen SH, Jacobsen LV, Petri KCC, Hale PM, Kordonouri O. Liraglutide in an Adolescent Population with Obesity: A Randomized, Double-Blind, Placebo-Controlled 5-Week Trial to Assess Safety, Tolerability, and Pharmacokinetics of Liraglutide in Adolescents Aged 12-17 Years. J Pediatr. 2017 Feb;181:146-153.e3. doi: 10.1016/j.jpeds.2016.10.076. Epub 2016 Dec 13. PMID 27979579
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com